CLINICAL TRIAL: NCT04267237
Title: A Phase II, Open-label, Multicenter, Randomized Study of the Efficacy and Safety of RO7198457 in Combination With Atezolizumab Versus Atezolizumab Alone Following Adjuvant Platinum-doublet Chemotherapy in Patients Who Are ctDNA Positive After Surgical Resection of Stage II-III Non-small Cell Lung Cancer
Brief Title: A Study of the Efficacy and Safety of RO7198457 in Combination With Atezolizumab Versus Atezolizumab Alone Following Adjuvant Platinum-Doublet Chemotherapy in Participants Who Are ctDNA Positive After Surgical Resection of Stage II-III Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Accrual timelines
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO41836; 2019-003449-14 (EudraCT Number)
Record Dates: First submitted 2020-02-07; First posted 2020-02-12 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: Cancer vaccine; Neoantigen; Personalized; Atezolizumab; Vaccine; Immunotherapy; Anti-PDL1; Checkpoint Inhibitor; Personalized vaccine; Non-small cell lung cancer; NSCLC; Adjuvant
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab

STUDY DESIGN:
Masking Description: Open label
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Atezolizumab (Experimental): Participants will receive atezolizumab on Day 1 of each 28-day cycle (Q4W) for 12 cycles.
  Interventions: Drug: Atezolizumab
- Atezolizumab + RO7198457 (Experimental): Participants will receive atezolizumab Q4W along with RO7198457 for 12 cycles.
  Interventions: Drug: Atezolizumab; Drug: RO7198457

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 1680 mg will be administered by intravenous (IV) infusion on Day 1 of Cycles 1-12.
  Other Names: Tecentriq
Drug: RO7198457 — RO7198457 will be administered by IV infusion at protocol-defined intervals for 12 cycles.
  Arms: Atezolizumab + RO7198457

SUMMARY:
This study will evaluate the efficacy, safety, pharmacokinetics, immunogenicity and biomarkers of RO7198457 plus atezolizumab compared with atezolizumab alone in patients with Stage II-III non-small cell lung cancer (NSCLC) who are circulating tumor DNA (ctDNA) positive following surgical resection and have received standard-of-care adjuvant platinum-doublet chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years;
* Resected Stage II-III Non-small Cell Lung Cancer (NSCLC) per American Joint Committee on Cancer staging criteria, 8th revised edition;
* Complete R0 resection of Stage II or III NSCLC prior to enrollment and adequate recovery from surgery;
* Pathological evaluation of mediastinal lymph nodes preoperatively or intraoperatively;
* ctDNA (circulating tumor DNA) identified in plasma after resection of Stage II-III NSCLC and prior to start of adjuvant platinum-doublet therapy, as determined by central testing;
* Treatment with at least two cycles of adjuvant platinum-doublet chemotherapy regimens for resected NSCLC;
* No unequivocal evidence of disease after surgery and adjuvant platinum-doublet chemotherapy, as assessed on imaging (computed tomography [CT] scan or magnetic resonance imaging [MRI]) within 28 days prior to randomization;
* Availability of adequate tumor material;
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1;
* Adequate hematologic and end-organ function;
* Negative HIV test at screening;
* Negative hepatitis B test at screening;
* Negative hepatitis C test at screening.

Exclusion Criteria:

* Participants with a known mutation in exons 18-21 of epidermal growth factor receptor (EGFR) or with a known anaplastic lymphoma kinase (ALK) or reactive oxygen species (ROS) alteration;
* History of malignancy other than disease under study within 5 years prior to enrollment, with the exception of malignancies with a negligible risk of metastasis or death, such as adequately treated carcinoma in situ of the cervix, non-melanoma skin cancer, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer;
* Induction and neoadjuvant systemic therapy prior to resection of NSCLC;
* Radiotherapy prior to or after resection of NSCLC;
* Prior systemic investigational therapy;
* Prior anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies, or a cancer vaccine;
* Treatment with systemic immunostimulatory agents within 6 weeks or 5 drug elimination half-lives, prior to initiation of study treatment;
* Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment or anticipation of need for systemic immunosuppressive medication during study treatment;
* Treatment with monoamine oxidase inhibitors (MAOIs) within 3 weeks prior to initiation of study treatment or requirement for ongoing treatment with MAOIs;
* Active or history of autoimmune disease or immune deficiency;
* Known primary immunodeficiencies, either cellular or combined T-cell and B-cell immunodeficiencies;
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan;
* Significant cardiovascular disease;
* Major surgical procedure, other than for diagnosis or for resection of disease under current study, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study;
* Known active or latent tuberculosis infection;
* Recent acute infection;
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during study treatment or within 5 months after the final dose of study treatment;
* Prior allogeneic stem cell or solid organ transplantation;
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the participants at high risk from treatment complications;
* Known clinically significant liver disease;
* Previous splenectomy;
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins;
* Known hypersensitivity to Chinese hamster ovary cell products or any component of the atezolizumab formulation;
* Known allergy or hypersensitivity to any component of RO7198457;
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-31 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival (DFS) | Up to 62 months
  DFS as assessed by the investigator, is defined as the time from randomization to the date of first documented recurrence of NSCLC or occurrence of new primary NSCLC or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) and Serious AEs (SAEs) determined according to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0) | Up to 90 days after the final dose of study drug or until initiation of another systemic anti-cancer therapy (up to approximately 62 months)
Plasma Concentrations of RNA at Specified Timepoints | Arm B: Days 1, 8, 15, 22 of Cycle 1 (each cycle is 28 days), Day 1 of Cycle 2, 3, 5, 7, 9, 11 and treatment discontinuation (TD) visit (up to 12 months)
Plasma Concentrations of (R)-N,N,N-trimethyl-2,3-dioleyloxy-1-propanaminium chloride (DOTMA) at Specified Timepoints | Arm B: Days 1, 8, 15, 22 of Cycle 1 (each cycle is 28 days), Day 1 of Cycle 2, 3, 5, 7, 9, 11 and treatment discontinuation (TD) visit (up to 12 months)
Maximum Serum Concentration (Cmax) of Atezolizumab at Specified Timepoints | Arm A and Arm B: Day 1 of Cycles 1-4 (each cycle is 28 days) and at TD visit (up to 12 months)
Minimum Serum Concentration (Cmin) of Atezolizumab at Specified Timepoints | Arm A and Arm B: Day 1 of Cycles 1-4 (each cycle is 28 days) and at TD visit (up to 12 months)
Change from Baseline in Number of Participants With Anti-drug Antibodies (ADA) to Atezolizumab | Arm A and Arm B: Baseline, Day 1 of Cycles 1-4 (each cycle is 28 days) and at TD visit (up to 12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform(www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).